CLINICAL TRIAL: NCT03245918
Title: Relative Bioavailability of an Extemporaneous Oral Suspension of Aprepitant in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lee Dupuis, Health Clinician Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000056100
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aprepitant Capsule Study Period #1 (Other)
  Interventions: Drug: Aprepitant Capsule 125 MG
- Aprepitant Oral Suspension Study Period#1 (Other)
  Interventions: Drug: Aprepitant oral suspension 20 mg/mL

INTERVENTIONS:
Drug: Aprepitant Capsule 125 MG — Patients will be randomized to either the aprepitant capsule or oral suspension for the first study period, and will receive the alternate formulation during the second study period
  Arms: Aprepitant Capsule Study Period #1
Drug: Aprepitant oral suspension 20 mg/mL — Patients will be randomized to either the aprepitant capsule or oral suspension for the first study period, and will receive the alternate formulation during the second study period
  Arms: Aprepitant Oral Suspension Study Period#1

SUMMARY:
Antiemetic therapies have improved in recent years, but chemotherapy-induced nausea and vomiting (CINV) are still common and are among the most distressing side effects of chemotherapy. Aprepitant is commercially available in Canada as capsules. An oral liquid aprepitant formulation would be ideal for oral administration to patients unable to swallow capsules.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by responsible physician (see 4.3) (i.e. have no clinically significant diseases captured in the medical history, on physical examination and/or laboratory tests)
* 18 to 55 years of age
* BMI within 18.5 to 30 kg/m2
* Non-smoker
* Systolic blood pressure between 90-140 mmHg, diastolic blood pressure between 60-90 mmHg, and heart rate between 60-100 bpm, inclusive.
* Female subjects of childbearing potential should be either sexually inactive (abstinent) or be using one of acceptable methods of birth control for 15 days prior to the first dose of the study, throughout the study and for at least 30 days after the last aprepitant dose.
* Able to swallow whole aprepitant capsules
* Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer.

Exclusion Criteria:

* Clinically significant illness or surgery within 8 weeks prior to dosing.
* Positive for hepatitis B, hepatitis C, or HIV at screening as per medical history.
* History of allergic reactions to the study drug and/or its excipients.
* Subjects concurrently treated with drugs that are metabolized through CYP3A4, including but not limited to pimozide, terfenadine, astemizole, or cisapride, ketoconazole, itraconazole, clarithromycin, diltiazem, warfarin, rifampin, carbamazepine, and phenytoin etc.
* History of drug or alcohol abuse within the last 6 months.
* Severe mental disorders.
* Blood donation of 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration.
* Pregnant or breastfeeding.
* Use of recreational drugs, prescription medications (other than hormonal contraceptive agents),non-prescription medications (over-the-counter) or natural health products within 7 days or 5 half-lives (whichever is longer) prior to the administration of the first dose of study medication.
* Consumed grapefruit or grapefruit products within 7 days of each study period
* Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability of the oral suspension relative to the capsule | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel P, Nathan PC, Walker SE, Zupanec S, Volpe J, Dupuis LL. Relative bioavailability of an extemporaneously prepared aprepitant oral suspension in healthy adults. J Oncol Pharm Pract. 2019 Dec;25(8):1907-1915. doi: 10.1177/1078155219828806. Epub 2019 Feb 5. PMID 31694495